CLINICAL TRIAL: NCT05944549
Title: Financial Coaching and Lifestyle Intervention for Diabetes Prevention in Low-income Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Bank of America Foundation (Unknown)
Responsible Party: Principal Investigator, Shreela V Sharma, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0002
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Weight Loss
Keywords: weight loss; financial coaching; Cognitive functioning; metabolic functioning; psychosocial measures; health behaviors
MeSH Terms: conditions — Weight Loss; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Intervention group (Experimental)
  Interventions: Behavioral: Financial coaching using TrustPlus; Behavioral: Brighter Bites; Behavioral: Noom
- lifestyle-intervention group (Active Comparator)
  Interventions: Behavioral: Brighter Bites; Behavioral: Noom

INTERVENTIONS:
Behavioral: Financial coaching using TrustPlus — Participants will be assigned a financial coach, who will, prepare a budget, conduct a soft pull of their credit report and score to analyze the credit score. Based on the participant's goals and financial limitations as highlighted by the, the participant and financial coach will create a personalized financial action plan comprising of strategies, follow-up actions, and resources, which includes unlimited access to one-on-one sessions with the financial coach. After the intensive financial coaching, participants will maintain access to the TrustPlus Portal and can continue to connect with their financial coach as needed throughout the 6-month intervention period. Participants will also have ongoing access to educational webinars and Trust+Ed, an interactive resource that provides self-guided content on many financial topics of interest, such as credit building and debt management.
  Arms: Enhanced Intervention group
Behavioral: Brighter Bites — Families receive a weekly distribution of fresh fruits and vegetables for 24 weeks, there will be Nutrition education in school throughout the school year using the evidence-based CATCH (Coordinated Approach to Child Health) program and weekly healthy recipe tastings and cooking skill demos for families during produce pick-up time.Fruit and vegetable access is complemented by CATCH, an evidence based, Texas Education Agency-approved, coordinated school health program designed to promote healthy nutrition, physical activity, and prevent obesity in schoolchildren. In addition, the Brighter Bites website and mobile app are freely available in English and Spanish.
Behavioral: Noom — Participants will get access to Noom which is a mobile app for weight loss that shifts the paradigm from dieting to a digitally supported and artificial intelligence (AI)-driven cognitive behavioral therapy approach to support personalized behavior changes towards eating, physical activity and stress management. The Noom Healthy Weight curriculum covers foundations in weight loss, nutrition, physical activity, sleep and stress management.Daily tasks (e.g., weight and food logs, readings) are organized vertically in simple cards on the phone screen, allowing users to easily scroll through what needs to be done. It will pull physical activity data (e.g., steps) directly from the health app on smartphones or apps associated with external devices such as Fitbit. Furthermore, Noom stands out from other app-based programs by assigning a personal coach to each user, helping users navigate the emotional and physiological experiences of the Noom weight loss experience.

SUMMARY:
The purpose of this study is to compare the effect on weight and metabolic outcomes of an enhanced intervention, comprised of evidence-based financial coaching plus a lifestyle intervention vs. the lifestyle intervention alone

ELIGIBILITY:
Inclusion Criteria:

* English speaking parents
* BMI>25.0 at baseline
* must have a child participant in the Brighter Bites program at study enrollment
* own a smartphone (Android 6 and iPhone 12.4 or later)
* must able to participate in study activities

Exclusion Criteria:

* medications known to affect appetite or body composition (e.g., corticosteroids, antidepressants, beta blockers, sulfonylureas, insulin)
* currently diagnosed with conditions known to affect body composition or fat distribution (e.g., Cushing's syndrome, hypothyroidism)
* diagnosis of an eating disorder
* currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Percent weight loss | From baseline to 3 months
  Average of the 2 weights will be calculated
Percent weight loss | From baseline to 6 months
  Average of the 2 weights will be calculated

SECONDARY OUTCOMES:
Change in cognitive functioning as assessed by the Flanker Inhibitory test for inhibitory control | Baseline, 3 months, 6 months
  The Flanker is a measure of executive function, specifically inhibitory control and attention. Total score ranges from 0-10, and a higher score indicates higher levels of ability to attend to relevant stimuli and inhibit attention from irrelevant stimuli.
Change in cognitive functioning as assessed by the List Sorting Working Memory Test for working memory | Baseline, 3 months, 6 months
  This test assesses working memory. Total score ranges from 0-26, with a higher score indicating better working memory.
Change in cognitive functioning as assessed by the Dimensional Change Card Sort Test (DCCS) for flexible shifting | Baseline, 3 months, 6 months
  The DCCS is a measure of cognitive flexibility. Total score ranges from 0-10, and a higher score indicates a higher level of cognitive flexibility.
Change in cognitive functioning as assessed by the Pattern Comparison Processing Speed Test for processing speed | Baseline, 3 months, 6 months
  This test measures speed of processing by asking participants to discern whether two side-by-side pictures are the same or not. Total score ranges from 0-130, with a higher score indicating greater processing speed.
Change in lipid levels | Baseline, 6 months
Change in HbA1C | Baseline, 6 months
Change in fasting plasma glucose (FPG) | Baseline, 6 months
Change in diastolic blood pressure | Baseline, 3 months, 6 months
Change in systolic blood pressure | Baseline, 3 months, 6 months
Change in financial Stress as assessed by the Financial Stress Questionnaire | Baseline, 3 months, 6 months
  Participants will be asked "Did any of the following happen to you because of a shortage of money in the past 6 months?," and participants will respond Yes or No to the following items. Data will be reported as the number of items for which participants answered "Yes"--total score ranges from 0-7, and a higher score indicates greater financial stress.
  Could not pay electricity, gas or telephone bills on time Could not pay the mortgage or rent on time Pawned or sold something Went without meals Was unable to heat home Asked for financial help from friends or family Asked for help from welfare/community organizations
Change in mental health as assessed by the Fast Track Project Financial Stress Questionnaire (affordability of household items) | Baseline, 3 months, 6 months
  This section of the questionnaire evaluates the affordability of 7 spending sources in the household (home, clothing, furniture, car, food, medical care and leisure) on a 1 to 5 scale (strongly agree, agree, neutral, disagree, strongly disagree). Total score ranges from 7 to 35, with a higher score indicating less affordability of household items.
Change in mental health as assessed by the Fast Track Project Financial Stress Questionnaire (difficulty paying bills) | Baseline, 3 months, 6 months
  This section of the questionnaire assesses how much difficulty participants had paying bills on a 1 to 5 scale (a great degree of difficulty to no difficulty at all), with a higher score indicating less difficulty paying bills.
Change in mental health as assessed by the Fast Track Project Financial Stress Questionnaire (money remaining at end of month) | Baseline, 3 months, 6 months
  This section of the questionnaire assesses how much money was left at the end of the month on a 1 to 4 scale (not enough, just enough, some money left, more than enough money left over), with a higher score indicating more money left at the end of the month.
Change in stress as assessed by the Perceived Stress Scale (PSS) | Baseline, 3 months, 6 months
  This is a 10 item questionnaire and each is scored from 0(never) to 4(very often) for a maximum score range of 0-40 a higher number indicating more stress
Change in anxiety as assessed by the Generalized Anxiety Disorder (GAD7) | Baseline, 3 months, 6 months
  This is a 7 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) for a maximum score range of 0-21 a higher number indicating more anxiety
Change in depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, 3 months, 6 months
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) for a maximum score range of 1-27 a higher number indicating more depression
Change in quality of life as assessed by the Center for Disease Control (CDC)Population Well-Being Survey | Baseline, 3 months, 6 months
  This is a 34-item questionnaire, and each item is scored on a 1-5 scale, with a higher value indicating greater well-being. Score on each of the 34 items will be reported in a separate row.
Change in quality of life as assessed by the Short-Form 12 (SF-12) | Baseline, 3 months, 6 months
  This is a 12 item questionnaire, scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Change in quality of life as assessed by the Subjective Happiness Scale (SHS) | Baseline, 3 months, 6 months
  This is a 4 item questionnaire and each is scored form 1-7, higher number indicating greater levels of happiness
Change in quality of life as assessed by the Satisfaction with Life Scale (SWLS) | Baseline, 3 months, 6 months
  This is a 5 item questionnaire and each is scored from 1( strongly disagree) to 7(strongly agree) for a maximum score range of 5-35, a higher number indicating better satisfaction
Change in health behaviors as assessed by the NCI Automated 24-hour Dietary Assessment (ASA24) to analyze diet patterns | Baseline, 3 months, 6 months
  This is a self reported outcome with support from a trained research dietitian by phone. ASA24 provides detailed information on intake of macronutrients and food groups, from which we can estimate the Healthy Eating Index,48 daily servings of fruit and vegetable intake, percent calorie intake from fat, protein and carbohydrates, and daily intake of sugar-sweetened beverages.
Change in physical activity as assessed by the School Physical Activity and Nutrition (SPAN) survey | Baseline, 3 months, 6 months
  Data will be reported in rows as the number of days per week that participants get the below amounts of exercise.
  Days per week of at least 60 min physical activity Days per week of at least 20 min vigorous physical activity Days per week of at least 30 min outdoor play
Change in sedentary behavior as assessed by the School Physical Activity and Nutrition (SPAN) survey | Baseline, 3 months, 6 months
  Data will be reported in rows as the number of hours per day that participants exhibit the below sedentary behaviors.
  Hours per day playing video games Hours per day watching Television or movies
Change in quality of sleep as assessed by the Pittsburgh Sleep Quality Index(PSQI) | Baseline, 3 months, 6 months
  This is a 19 item questionnaire. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Change in food security as assessed by the National Health Interview Survey(NHIS) Food Insecurity Screener | Baseline, 3 months, 6 months
  This is a 10 item questionnaire and the first 3 questions are scored from 1(often true) to 3(never true),the fifth and 10 questions are scored from 1(almost every month) to 3(only 1 or 2 months) and all other questions are answered as yes or no.
  Responses of "yes," "often," "sometimes," "almost every month," and "some months but not every month" were defined as affirmative responses. Based on the summed number of affirmative answers, food security was categorized into four levels: high food security (0 item affirmed), marginal food security (1-2 items affirmed), low food security (3-5 items affirmed), and very low food security (6-10 items affirmed). Participants with low or very low food security were considered food insecure.

CONTACTS AND LOCATIONS:
Overall Officials: Shreela V Sharma, PhD,RD,LD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No